CLINICAL TRIAL: NCT06348641
Title: The Effect of Massage Applied Before The Retinopathy of Prematurity Examination on the Pain Level and Comfort of the Newborn
Brief Title: Reducing Pain and Increasing Comfort During a Retinopathy of Prematurity Examination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nurgül Tekin (Other)
Responsible Party: Sponsor-Investigator, Nurgül Tekin, Principal Investigator, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-KAEK-25 2022/12-11
Record Dates: First submitted 2024-03-10; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Pain; Retinopathy of Prematurity; Premature Baby 26 to 32 Weeks; Premature Baby 33 to 36 Weeks
MeSH Terms: conditions — Pain; Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: In the calculation of the sample size, the power level was 80% and the significance level was 5%. When the effect size was determined as 0.8 in the examination of the difference between the experimental and control groups in terms of the premature infant pain profile (PIPP) variable, it was determined by the statistical expert that the number of babies to be included in each group was 26 and 52 babies in total should be included in the study. Based on this, the study sample was determined as 60 preterm infants in 30 experimental and 30 control groups. Block randomization method will be applied in the randomization of the groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Babies in intervention classes will receive baby massage before the examination. Pre-examination baby massage will be applied by a single nurse = researcher. Video recording will be taken before and during the ROP examination, and evaluations will be made by two neonatal nurses other than the researcher.
  Babies will be massaged by the researcher in accordance with IAIM rules and massage techniques. The total massage time will be equal for each baby.
  Interventions: Other: baby massage
- control group (No Intervention): For the control group, the routine retinopathy examination of the unit will be performed without any intervention.
  Video recording will be taken before and during the ROP examination, and evaluations will be made by two neonatal nurses other than the researcher.

INTERVENTIONS:
Other: baby massage — The infant massage to be applied before the examination will be applied by a single nurse=researcher. Video recordings will be taken before and during the ROP examination and evaluations will be made by two neonatal nurses other than the researcher.
  Arms: experimental group

SUMMARY:
The aim of this study is to investigate the effect of baby massage applied to babies with retinopathy of prematurity on the pain and comfort of the newborn.

This was randomised-controlled study in the NICU at the Health Sciences University Bursa High Specialization Training and Research Hospital, Bursa, Turkey. The population of the study will consist of preterms hospitalized in the neonatal intensive care unit during the time period of the study. In the calculation of the sample size, the power level was 80% and the significance level was 5%. When the effect size was determined as 0.8 in the examination of the difference between the experimental and control groups in terms of the premature infant pain profile (PIPP) variable, it was determined by the statistical expert that the number of babies to be included in each group was 26 and 52 babies in total should be included in the study. Based on this, the study sample was determined as 60 preterm infants in 30 experimental and 30 control groups. Block randomization method will be applied in the randomization of the groups.

Case report form, PIPP=Premature Infant Pain Scale and Premature Infant Comfort Scale (PBIQ) will be used to collect the study data. Patients included in the study will be examined by the same ophthalmologist.

The infant massage to be applied before the examination will be applied by a single nurse=researcher. Video recordings will be taken before and during the ROP examination and evaluations will be made by two neonatal nurses other than the researcher.

Infants will be massaged by the researcher in accordance with IAIM guidelines and massage techniques. Total massage time will be equal for each infant.

The researcher has an IAIM infant massage certificate. Before starting the infant massage, jewelry will be removed and hands will be washed. In the study, leg and face massage will be applied among the massage techniques in the IAIM guidelines.

ELIGIBILITY:
Inclusion Criteria:

* <32 gestational age
* Birth weight of <1500g
* Who were clinical stable
* Baby's first eye examination
* The baby's family has permission

Exclusion Criteria:

* Infants with previous ROP examination
* Lack of mechanical ventilator support
* Major congenital anomaly
* Intraventriculer bleeding
* Receiving analgesic medication

Ages: 1 Day to 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Pain during examination for retinopathy of prematurity | Before, during and after ROP examination
  Reducing the premature baby pain scale score of the experimental group compared to the control group.
  It is suitable for term and preterm babies and is used to evaluate acute and procedural pain. Scoring ranges from 0 to 21, with a score of six or lower being considered as no or minimal pain, between 7-12 points as moderate pain, and between 13-21 points as severe pain. It is evaluated 15 seconds before the intervention and 30 seconds after the intervention.

SECONDARY OUTCOMES:
Comfort during retinopathy of prematurity examination | Before, during and after ROP examination
  Reducing the premature baby comfort scale score of the experimental group compared to the control group.
  It is a multidimensional scale used to evaluate behavioral and psychological comfort and pain. Premature baby comfort scale evaluates 7 parameters such as Alertness, Calm/Agitation, Respiratory Status (only in mechanical ventilation support) or Crying (not evaluated because it is scored only in children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate. Each item is a 5-point Likert type, scored from 1 to 5, from worst to best.
  According to the scale, 35 indicates the lowest and 7 indicates the highest comfort score. A high score from the scale indicates that the comfort level is low. If the total score obtained is ≥17, it is the cut-off value of the scale, it is the limit value for the baby's comfort level and indicates the need for a pain-reducing intervention.

IPD SHARING:
Plan to Share IPD: No